CLINICAL TRIAL: NCT02645747
Title: RETRO CRVO: Retrospective Data Analysis of Patients Treated for Macular Edema Due to Central Retinal Vein Occlusion
Brief Title: Retrospective Data Analysis of Patients Treated for Macular Edema Due to Central Retinal Vein Occlusion
Acronym: RETRO CRVO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 18586
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: The source population of this study is patients who suffer from visual impairment due to ME secondary to CRVO. In order to ensure the representativeness of the study population, the number of Belgian patients which started Eylea treatment during the brief period between the 1st of June 2014 and the 28th of February 2015 were taken into account. However, data of patients diagnosed with neovascular glaucoma secondary to CRVO will be excluded.
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — Eylea (intravitreal aflibercept) is an anti-Vascular Endothelial Growth Factor (VEGF) drug indicated for neovascular age-related macular degeneration (AMD), visual impairment due to diabetic macular edema (DME) and visual impairment due to macular edema (ME) secondary to central or branched retinal vein occlusion (RVO).
  RVO, both branch and central, is the second most common type of retinal vascular disorders after diabetic retinal disease. Central retinal vein occlusion (CRVO) is characterized by an obstruction of the central retinal vein combined with variable amounts of retinal arterial insufficiency.

SUMMARY:
The objective of this retrospective chart review is to evaluate drug utilization, usage patterns and indication of effectiveness Eylea in the routine clinical (real-life) management of patients who suffer from ME (Macular Edema), secondary to CRVO (Central Retinal Vein Occlusion), and who started treatment with Eylea for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients who suffer from visual impairment due to ME secondary to CRVO
* Anti-VEGF treatment-naive patients who started reimbursed Eylea treatment between the 1st of June 2014 and the 28th of February 2015

Exclusion Criteria:

* Patients diagnosed with neovascular glaucoma secondary to CRVO will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population of this study is patients who suffer from visual impairment due to macular edema secondary to central retinal vein occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Treatment duration | At 12 months of treatment with Eylea
Number of eyes treated (mono-and biocular) | At 12 months of treatment with Eylea
Change in visual acuity (BCVA score) | At 12 months of treatment with Eylea
Number of Eylea injections per treated eye | At 12 months of treatment with Eylea

SECONDARY OUTCOMES:
Estimation of percentage (%) of eyes which need additional treatment after 2 years at the discretion of the treating physician. | At 12 months of treatment with Eylea
Sufficiency of reimbursed number of Eylea injections (max. 9 injections/eye in year 1) for treatment of all patients during the first year of treatment. | At 12 months of treatment with Eylea
Number of patients who discontinued their treatment with Eylea prematurely | At 12 months of treatment with Eylea
  Investigator is asked to categorize the number of patients who ended their treatment prematurely according to the following reasons :
  * Lost-to-follow up (measured as number of patients)
  * Lack of efficacy (measured as number of patients)
  * Remission (measured as number of patients)
  * AE (measured as number of patients)
  * Other (measured as number of patients)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Belgium